CLINICAL TRIAL: NCT05966090
Title: A Phase III, Open-label, Randomized, Controlled, Multi-country Study to Evaluate the Immune Response, Safety and Reactogenicity of RSVPreF3 OA Investigational Vaccine When Co-administered With Herpes Zoster Recombinant Subunit (HZ/su) Vaccine in Adults Aged 50 Years and Older
Brief Title: A Study on Safety and Immune Response of Investigational RSV OA Vaccine in Combination With Herpes Zoster Vaccine in Healthy Adults
Acronym: RSV-OA=ADJ-020
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 219331
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Syncytial Viruses; Respiratory Syncytial Virus Infections
Keywords: Respiratory syncytial virus; Infection; Vaccine; Older adult; Immunogenicity; Safety
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Co-administration Group (Experimental): Participants received both herpes zoster recombinant subunit (HZ/su) vaccine and respiratory syncytial virus prefusion protein 3 older adult (RSVPreF3 OA) vaccine on Day 1 followed by second dose of HZ/su vaccine on Day 61.
  Interventions: Biological: RSVPreF3 OA investigational vaccine; Biological: HZ/su vaccine
- Control Group (Active Comparator): Participants received HZ/su vaccine on Day 1 and RSVPreF3 OA vaccine on Day 31 followed by second dose of HZ/su vaccine on Day 61.
  Interventions: Biological: RSVPreF3 OA investigational vaccine; Biological: HZ/su vaccine

INTERVENTIONS:
Biological: RSVPreF3 OA investigational vaccine — One dose of RSVPreF3 OA investigational vaccine given intramuscularly on Day 1 (Coadministration group) or Day 31 (Control group).
  Other Names: Respiratory Syncytial Virus PreFusion protein 3 Older Adults vaccine
Biological: HZ/su vaccine — Two doses of HZ/su vaccine given intramuscularly on Day 1 and Day 61.
  Other Names: Herpes Zoster recombinant subunit vaccine, Shingrix

SUMMARY:
To assess the ability of RSVPreF3 OA investigational vaccine to generate an immune response when given in combination with HZ/su vaccine and its safety in older adults, aged >=50 years of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female participant ≥50 YOA at the time of the first study intervention administration.
* Female participants of non-childbearing potential may be enrolled in the study.
* Female participants of childbearing potential may be enrolled in the study, if the participant:

  * has practiced adequate contraception from 1 month prior to study intervention administration.
  * has a negative pregnancy test on the day of and prior to study intervention administration.
  * has agreed to continue effective contraception until the end of the study.
* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol. Written or witnessed informed consent obtained from the participant prior to any study specific procedure being performed.
* Participants living in the general community or in an assisted-living facility that provides minimal assistance, such that the participant is primarily responsible for self-care and activities of daily living.
* Participants who are medically stable in the opinion of the investigator at the time of first study intervention administration. Participants with chronic stable medical conditions with or without specific treatment, such as diabetes mellitus, hypertension, or cardiac disease, are allowed to participate in this study if considered by the investigator as medically stable.

Exclusion Criteria:

* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any confirmed or suspected autoimmune disorders, immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions, in particular any history of severe allergic reaction to any vaccine component.
* History of Guillain-Barré syndrome.
* Any history of dementia or any medical condition that moderately or severely impairs cognition.
* Recurrent or uncontrolled neurological disorders or seizures. Participants with medically controlled chronic neurological diseases can be enrolled in the study as per investigator assessment, provided that their condition will allow them to comply with the requirements of the protocol.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Clinically suspected or polymerase chain reaction (PCR)-confirmed ongoing episode of herpes zoster.
* History of previous vaccination with any licensed or investigational recombinant adjuvanted zoster vaccine (HZ/su vaccine; Shingrix) before the study start or planned receipt through study participation.
* History of previous vaccination with any licensed or investigational live herpes zoster vaccine (Zostavax) in the last 2 years from enrollment, or planned receipt through study participation.
* Previous vaccination with licensed or investigational RSV vaccine.
* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study interventions during the period beginning 30 days before the first dose of study interventions, or their planned use during the study period.
* Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first study intervention administration and ending 30 days after the last study intervention administration.

  o In the case of COVID-19 and inactivated/subunit/split influenza vaccines, this time window can be decreased to 14 days before and after each study intervention administration provided COVID-19 vaccine use is in line with local governmental recommendations.
* Planned or actual administration of adjuvanted quadrivalent influenza vaccine influenza vaccine not foreseen by the study protocol in the period starting 30 days before the first study intervention administration and ending 30 days after the last study intervention administration.
* Administration of long-acting immune-modifying drugs during the period starting 180 days before the administration of first dose of study interventions or planned administration at any time during the study period (e.g., infliximab).
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the administration of first dose of study interventions or planned administration during the study period.
* Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune modifying drugs during the period starting 90 days prior to the first study intervention dose or planned administration during the study period. For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent. Inhaled, topical or intra-articular steroids are allowed.
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non investigational vaccine/product (IMP) (drug or invasive medical device).
* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.Bedridden participants.
* Planned move during the study conduct that prohibits participation until study end.
* Participation of any study personnel or their immediate dependents, family, or household members.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-07-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (11):
  - GSK Investigational Site, Daphne, Alabama
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Corte Madera, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, North Miami Beach, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Versailles, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, San Antonio, Texas
- Canada (11):
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Guelph, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Brampton
  - GSK Investigational Site, Guelph
  - GSK Investigational Site, Québec
  - GSK Investigational Site, Sarnia
  - GSK Investigational Site, Sherbrooke
  - GSK Investigational Site, Toronto

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in adult participants aged 50 years and older, in 20 study sites.
Pre-assignment Details: A total of 530 eligible participants were randomized in a 1:1 ratio to either co-administration group or control group at Day 1.
Period: Overall Study
Arm/Group | Co-administration Group | Control Group
Started | 265 | 265
Completed | 256 | 255
Not Completed | 9 | 10
Not completed — Lost to Follow-up | 6 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol-Specified Withdrawal Criterion Met | 0 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Exposed set included all participants in the enrolled set who received at least 1 study intervention.
Groups:
- Co-administration Group: Participants received both HZ/su vaccine and RSVPreF3 OA vaccine on Day 1 followed by second dose of HZ/su vaccine on Day 61.
- Total: Total of all reporting groups
Arm/Group | Co-administration Group | Control Group | Total
Number analyzed (Participants) | 265 | 265 | 530
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (8.56) | 63.9 (8.73) | 63.9 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 146 | 292
  Male | 119 | 119 | 238
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 30 | 58
  Not Hispanic or Latino | 237 | 235 | 472
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Geometric Mean Concentration (GMC) of Anti-glycoprotein E (gE) Antibodies at 1 Month Post-second Dose of HZ/su Vaccination
Description: Anti-gE antibodies were measured with enzyme linked immunosorbent assay (ELISA) and the results were expressed as GMC, in milli international units per milliliter (mIU/mL).
Time Frame: At 1 month post-second dose of HZ/su vaccination (Day 91)
Population: Per protocol set for HZ/su included all eligible participants in the exposed set who: received 2 doses of HZ/su vaccine, had immunogenicity results for anti-gE antibody concentrations, complied with the blood draw interval, without intercurrent medical conditions and without prohibited concomitant medication/vaccination, did not met any of the criteria for elimination up to blood sample collection. Participants with data available at the time of analysis were reported in this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 199 | 168
mIU/mL | 49326.9 [44948.5 to 54131.7] | 61192.7 [55306.4 to 67705.5]
Statistical Analysis 1: Comparison: Co-administration Group vs Control Group; To demonstrate non-inferiority of the humoral immune response to 2 doses of HZ/su vaccine when the first dose of HZ/su vaccine was co-administered with RSVPreF3 OA investigational vaccine, compared to 2 doses of HZ/su vaccine administered alone; Test type: Non-Inferiority — Non - Inferiority (NI) was to be demonstrated if the upper limit of the 2 sided 95% confidence interval (CI) of the GMC ratio between the Control group (at Day 91) versus Co-administration group (at Day 91) for anti-gE Ab 1-month after the second HZ/su vaccine dose was <=1.5; Ratio = 1.24, 95% CI 2-sided [1.08 to 1.42] — The analysis of covariance (ANCOVA) model, for logarithm-transformed concentration, included the treatment group and age category at vaccination as fixed effects and the pre-dose log-10 titer as a covariate

2. Primary Outcome: Adjusted Geometric Mean Titers (GMT) of Respiratory Syncytial Virus-A (RSV-A) Neutralizing Titers [Estimated Dilution 60 (ED60)] at 1 Month After the RSVPreF3 OA Vaccination
Description: Neutralizing titers were measured with neutralization assay and the results were expressed as GMT. The ED60 was defined as the dose that produced an effect in 60% of the population.
Time Frame: At Day 31 for Co-administration Group and at Day 61 for Control Group
Population: Per protocol set for RSVPreF3 OA included all eligible participants in the exposed set who: received the RSVPreF3 OA vaccine, had immunogenicity results for RSV neutralizing titers, complied with the blood draw interval, without intercurrent medical conditions and without prohibited concomitant medication/vaccination and who did not met any of the criteria for elimination up to blood sample collection.Participants with data available at the time of analysis were reported in this outcome measure
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 237 | 218
Titers | 8426.8 [7504.2 to 9462.7] | 9628.7 [8532.7 to 10865.4]
Statistical Analysis 1: Comparison: Co-administration Group vs Control Group; To demonstrate the non-inferiority of RSVPreF3 OA investigational vaccine when co-administered with the first dose of HZ/su vaccine, compared to RSVPreF3 OA investigational vaccine administered alone; Test type: Non-Inferiority — NI was to be demonstrated if upper limit of the 2 sided 95% CI of the GMT ratio between the Control group (at Day 61) versus Co-administration group (at Day 31) for RSV-A neutralizing titer 1-month after the RSVPreF3 OA investigational vaccine dose was <=1.5; ratio = 1.14, 95% CI 2-sided [0.97 to 1.35] — The ANCOVA model, for logarithm-transformed titers, included the treatment group and age category at vaccination as fixed effects and the pre-dose log-10 titer as a covariate

3. Primary Outcome: Adjusted GMTs of RSV-B Neutralizing Titers (ED60) at 1 Month After the RSVPreF3 OA Vaccination
Description: as for outcome 2
Time Frame: At Day 31 for Co-administration Group and at Day 61 for Control Group
Population: Per protocol set for RSVPreF3 OA. Participants with data available at the time of analysis were reported in this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 237 | 218
Titers | 10354.2 [9288.4 to 11542.3] | 10143.4 [9057.5 to 11359.4]
Statistical Analysis 1: Comparison: Co-administration Group vs Control Group; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — NI was to be demonstrated if the upper limit of the 2 sided 95% CI of the GMT ratio between the Control group (at Day 61) versus Co-administration group (at Day 31) for RSV-B neutralizing titer 1-month after the RSVPreF3 OA investigational vaccine dose was <=1.5; ratio = 0.98, 95% CI 2-sided [0.84 to 1.15] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants With Seropositivity at Pre-vaccination and 1 Month Post-second Dose of HZ/su Vaccination
Description: Seropositivity was defined as the percentage of participants whose antibody concentration was greater than or equal to the assay cut-off value (97 mIU/mL).
Time Frame: Pre-vaccination (Day 1) and 1 month post-second dose of HZ/su vaccination (Day 91)
Population: Per protocol set for HZ/su. Only those participants with available data at specified timepoints were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 261 | 262
Percentage of participants
  Pre-vaccination (Day 1) | 98.5 [96.1 to 99.6] | 97.3 [94.6 to 98.9]
  1 month post-second dose of HZ/su vaccination (Day 91): number analyzed (Participants) | 198 | 170
  1 month post-second dose of HZ/su vaccination (Day 91) | 100.0 [98.2 to 100.0] | 100.0 [97.9 to 100.0]

5. Secondary Outcome: GMC of Anti-glycoprotein Antibodies at Pre-vaccination and 1 Month Post-second Dose of HZ/su Vaccination
Description: Anti-gE antibodies were measured with ELISA and the results were expressed as GMC.
Time Frame: Pre-vaccination (Day 1) and 1 month post-second dose of HZ/su vaccination (Day 91)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 261 | 262
mIU/mL
  Pre-vaccination (Day 1) | 1739.4 [1503.4 to 2012.5] | 1492.2 [1278.5 to 1741.5]
  1 month post-second dose of HZ/su vaccination (Day 91): number analyzed (Participants) | 198 | 170
  1 month post-second dose of HZ/su vaccination (Day 91) | 50235.2 [46013.4 to 54844.4] | 61204.7 [54959.6 to 68159.4]

6. Secondary Outcome: Mean Geometric Increase (MGI) of Anti-glycoprotein Antibodies at Pre-vaccination and 1 Month Post-second Dose of HZ/su Vaccination
Description: The MGI was defined as the geometric mean of the within participant ratios of the post-vaccination titer over the pre-vaccination titer. Anti-gE antibodies were measured with ELISA.
Time Frame: At 1 month post-second dose of HZ/su vaccination (Day 91) compared to Pre-vaccination (Day 1)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 198 | 170
Ratio | 28.24 [23.66 to 33.71] | 43.24 [34.97 to 53.47]

7. Secondary Outcome: Vaccine Response Rate (VRR) at 1 Month Post-second Dose of HZ/su Vaccination
Description: The VRR was defined as the percentage of participants who had at least: a 4-fold increase post-vaccination anti-gE antibody concentration as compared to (over) the pre-vaccination anti-gE antibody concentration (for participants who were seropositive at pre-vaccination); or, a 4-fold increase post-vaccination anti-gE antibody concentration as compared to (over) the anti-gE antibody cut-off value for seropositivity (97 mIU/mL) (for participants who were seronegative at pre-vaccination).
Time Frame: At 1 month post-second dose of HZ/su vaccination (Day 91)
Population: Per protocol set for HZ/su. Only those participants with available data at specified timepoint were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 198 | 170
Percentage of participants | 92.9 [88.4 to 96.1] | 96.5 [92.5 to 98.7]

8. Secondary Outcome: GMT of RSV-A Neutralizing Titers (ED60) at Pre-vaccination and 1 Month After the RSVPreF3 OA Vaccination
Description: as for outcome 2
Time Frame: At pre-vaccination (Day 1) and Day 31 for Co-administration Group and at pre-vaccination (Day 1) and Day 61 for Control Group
Population: Per protocol set for RSVPreF3 OA. Only those participants with available data at specified timepoints were included in this analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 261 | 249
Titers
  Pre-vaccination (Day 1) | 1005.4 [909.1 to 1111.9] | 961.2 [860.8 to 1073.4]
  Day 31: number analyzed (Participants) | 247 | 0
  Day 31 | 8553.3 [7568.7 to 9666.1] |
  Day 61: number analyzed (Participants) | 0 | 219
  Day 61 |  | 9689.4 [8561.7 to 10965.7]

9. Secondary Outcome: MGI of Respiratory Syncytial Virus-A Neutralizing Titers at 1 Month After the RSVPreF3 OA Vaccination
Description: The MGI was defined as the geometric mean of the within participant ratios of the post-vaccination titer over the pre-vaccination titer. Neutralizing titers were measured with neutralization assay.
Time Frame: At 1 month after the RSVPreF3 OA vaccine dose (Day 31 for Co-administration Group and Day 61 for Control Group) compared to Pre-vaccination (Day 1 for Co-administration Group and Control Group)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 247 | 219
Ratio | 8.55 [7.44 to 9.82] | 9.91 [8.55 to 11.49]

10. Secondary Outcome: GMT of RSV-B Neutralizing Titers (ED60) at Pre-vaccination and 1 Month After the RSVPreF3 OA Vaccination
Description: as for outcome 2
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 261 | 249
Titers
  Pre-vaccination (Day 1) | 1148.8 [1042.2 to 1266.3] | 1167.9 [1033.5 to 1319.8]
  Day 31: number analyzed (Participants) | 247 | 0
  Day 31 | 10521.3 [9411.3 to 11762.2] |
  Day 61: number analyzed (Participants) | 0 | 219
  Day 61 |  | 10352.2 [9122.8 to 11747.3]

11. Secondary Outcome: MGI of RSV-B Neutralizing Titers at 1 Month After the RSVPreF3 OA Vaccination
Description: as for outcome 9
Time Frame: as for outcome 9
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 247 | 219
Ratio | 9.01 [7.93 to 10.24] | 8.69 [7.50 to 10.07]

12. Secondary Outcome: Percentage of Participants With Solicited Administration Site Adverse Events (AEs) After Each Vaccine Dose Administration
Description: The solicited administration site events after vaccination included pain, erythema/redness, and swelling.
Time Frame: Within 7 days (the day of vaccination and 6 subsequent days) after each vaccine administration (vaccines administered at Days 1 and 61 for Co-Administration Group and at Days 1, 31 and 61 for Control group)
Population: Exposed set included all participants in the enrolled set who received at least 1 study intervention. Only those participants with solicited AEs were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 253 | 251
Percentage of participants
  Pain at injection site, HZ/su dose 1, given at Day 1 | 67.6 [61.4 to 73.3] | 59.8 [53.4 to 65.9]
  Pain at injection site, RSV dose, given at Day 1: number analyzed (Participants) | 252 | 0
  Pain at injection site, RSV dose, given at Day 1 | 63.1 [56.8 to 69.1] |
  Pain at injection site, RSV dose, given at Day 31: number analyzed (Participants) | 0 | 236
  Pain at injection site, RSV dose, given at Day 31 |  | 49.6 [43.0 to 56.1]
  Pain at injection site, HZ/su dose 2, given at Day 61: number analyzed (Participants) | 225 | 235
  Pain at injection site, HZ/su dose 2, given at Day 61 | 57.3 [50.6 to 63.9] | 63.4 [56.9 to 69.6]
  Erythema at injection site, HZ/su dose 1, given at Day 1 | 14.6 [10.5 to 19.6] | 13.1 [9.2 to 18.0]
  Erythema at injection site, RSV dose, given at Day 1: number analyzed (Participants) | 252 | 0
  Erythema at injection site, RSV dose, given at Day 1 | 7.9 [4.9 to 12.0] |
  Erythema at injection site, RSV dose, given at Day 31: number analyzed (Participants) | 0 | 236
  Erythema at injection site, RSV dose, given at Day 31 |  | 7.6 [4.6 to 11.8]
  Erythema at injection site, HZ/su dose 2, given at Day 61: number analyzed (Participants) | 225 | 235
  Erythema at injection site, HZ/su dose 2, given at Day 61 | 16.0 [11.5 to 21.5] | 11.9 [8.1 to 16.8]
  Swelling at injection site, HZ/su dose 1, given at Day 1 | 8.7 [5.5 to 12.9] | 8.8 [5.6 to 13.0]
  Swelling at injection site, RSV dose, given at Day 1: number analyzed (Participants) | 252 | 0
  Swelling at injection site, RSV dose, given at Day 1 | 6.0 [3.4 to 9.6] |
  Swelling at injection site, RSV dose, given at Day 31: number analyzed (Participants) | 0 | 236
  Swelling at injection site, RSV dose, given at Day 31 |  | 5.5 [3.0 to 9.2]
  Swelling at injection site, HZ/su dose 2, given at Day 61: number analyzed (Participants) | 225 | 235
  Swelling at injection site, HZ/su dose 2, given at Day 61 | 8.9 [5.5 to 13.4] | 8.5 [5.3 to 12.8]

13. Secondary Outcome: Percentage of Participants With Solicited Systemic AEs After Each Vaccine Dose Administration
Description: The solicited systemic events after vaccination included arthralgia, fatigue, fever (pyrexia), headache, myalgia, shivering/chills, and gastrointestinal symptoms (nausea, vomiting, diarrhea, and abdominal pain).
Time Frame: as for outcome 12
Population: Exposed set. Only those participants with solicited AEs were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 258 | 260
Percentage of participants
  Fever, Dosing at Day 1 | 8.9 [5.7 to 13.1] | 6.2 [3.6 to 9.8]
  Fever, Dosing at Day 31: number analyzed (Participants) | 0 | 245
  Fever, Dosing at Day 31 |  | 3.3 [1.4 to 6.3]
  Fever, Dosing at Day 61: number analyzed (Participants) | 230 | 243
  Fever, Dosing at Day 61 | 3.0 [1.2 to 6.2] | 7.4 [4.4 to 11.5]
  Headache, Dosing at Day 1 | 37.2 [31.3 to 43.4] | 30.0 [24.5 to 36.0]
  Headache, Dosing at Day 31: number analyzed (Participants) | 0 | 245
  Headache, Dosing at Day 31 |  | 22.9 [17.8 to 28.6]
  Headache, Dosing at Day 61: number analyzed (Participants) | 230 | 243
  Headache, Dosing at Day 61 | 30.9 [25.0 to 37.3] | 33.3 [27.4 to 39.6]
  Fatigue, Dosing at Day 1 | 48.8 [42.6 to 55.1] | 36.2 [30.3 to 42.3]
  Fatigue, Dosing at Day 31: number analyzed (Participants) | 0 | 245
  Fatigue, Dosing at Day 31 |  | 31.8 [26.1 to 38.1]
  Fatigue, Dosing at Day 61: number analyzed (Participants) | 230 | 243
  Fatigue, Dosing at Day 61 | 39.6 [33.2 to 46.2] | 46.5 [40.1 to 53.0]
  Myalgia, Dosing at Day 1 | 51.9 [45.7 to 58.2] | 40.4 [34.4 to 46.6]
  Myalgia, Dosing at Day 31: number analyzed (Participants) | 0 | 245
  Myalgia, Dosing at Day 31 |  | 26.9 [21.5 to 33.0]
  Myalgia, Dosing at Day 61: number analyzed (Participants) | 230 | 243
  Myalgia, Dosing at Day 61 | 37.0 [30.7 to 43.5] | 41.6 [35.3 to 48.0]
  Arthralgia, Dosing at Day 1 | 24.0 [18.9 to 29.7] | 16.2 [11.9 to 21.2]
  Arthralgia, Dosing at Day 31: number analyzed (Participants) | 0 | 245
  Arthralgia, Dosing at Day 31 |  | 12.7 [8.8 to 17.5]
  Arthralgia, Dosing at Day 61: number analyzed (Participants) | 230 | 243
  Arthralgia, Dosing at Day 61 | 20.9 [15.8 to 26.7] | 21.0 [16.0 to 26.7]
  Chills, Dosing at Day 1 | 22.9 [17.9 to 28.5] | 12.7 [8.9 to 17.4]
  Chills, Dosing at Day 31: number analyzed (Participants) | 0 | 245
  Chills, Dosing at Day 31 |  | 13.1 [9.1 to 17.9]
  Chills, Dosing at Day 61: number analyzed (Participants) | 230 | 243
  Chills, Dosing at Day 61 | 23.0 [17.8 to 29.0] | 25.9 [20.5 to 31.9]
  Gastrointestinal Symptoms, Dosing at Day 1 | 15.9 [11.7 to 20.9] | 15.0 [10.9 to 19.9]
  Gastrointestinal Symptoms, Dosing at Day 31: number analyzed (Participants) | 0 | 245
  Gastrointestinal Symptoms, Dosing at Day 31 |  | 11.4 [7.7 to 16.1]
  Gastrointestinal Symptoms, Dosing at Day 61: number analyzed (Participants) | 230 | 243
  Gastrointestinal Symptoms, Dosing at Day 61 | 9.1 [5.7 to 13.6] | 12.3 [8.5 to 17.2]

14. Secondary Outcome: Percentage of Participants With Unsolicited Adverse Events
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study vaccine, which does not necessarily have a causal relationship with study vaccine. An unsolicited AE was an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events. Unsolicited AEs must had been communicated by participant/participant's caregiver(s) who had signed the informed consent. Unsolicited AEs included both serious and non-serious AEs.
Time Frame: Within 30 days (the day of vaccination and 29 subsequent days) after vaccine administration
Population: Exposed set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 265 | 265
Percentage of participants | 23.4 [18.4 to 29.0] | 30.2 [24.7 to 36.1]

15. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: An SAE was defined as any untoward medical occurrence that, at any dose, resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event.
Time Frame: From first dose of study vaccine administration (Day 1) up to 6 months after last dose of study vaccine administration, approximately 241 days
Population: Exposed set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 265 | 265
Percentage of participants | 4.9 [2.6 to 8.2] | 2.3 [0.8 to 4.9]

16. Secondary Outcome: Percentage of Participants With Potential Immune-mediated Diseases (pIMDs)
Description: The pIMD was a subset of adverse events of special interest that included autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: as for outcome 15
Population: Exposed set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 265 | 265
Percentage of participants | 0.4 [0.0 to 2.1] | 0.8 [0.1 to 2.7]

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected up to Day 7 post each vaccination. Unsolicited AEs were collected up to Day 30 post each vaccination. SAEs and pIMDs were collected throughout the study period from Day 1 up to 6 months post last vaccination (approximately up to 241 days).
Description: Solicited and unsolicited events were reported per participant at any dose for the assessed timeframe (within 30 days after any vaccine dose administration) according to occurrence of each event, as pre-specified in Statistical Analysis Plan.
Arm/Group | Co-administration Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/265 | 0/265
Serious Adverse Events (participants affected / at risk) | 13/265 | 6/265
Other Adverse Events (participants affected / at risk) | 240/265 | 235/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-administration Group (N=265) | Control Group (N=265)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-administration Group (N=265) | Control Group (N=265)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 2 (2) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (2)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 23 (24) | 26 (31)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 30 (33) | 43 (56)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 149 (213) | 156 (232)
Influenza like illness (General disorders) | 1 (1) | 5 (5)
Injection site bruising (General disorders) | 0 (0) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (2) | 0 (0)
Injection site lymphadenopathy (General disorders) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 1 (1) | 2 (2)
Injection site warmth (General disorders) | 0 (0) | 1 (3)
Vaccination site reaction (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergy to vaccine (Immune system disorders) | 0 (0) | 2 (2)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 11 (11) | 11 (11)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (8) | 6 (7)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bladder injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Body temperature decreased (Investigations) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 1 (1) | 0 (0)
Troponin T increased (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 86 (112) | 78 (107)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 2 (3) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 27 (30) | 34 (40)
Vomiting (Gastrointestinal disorders) | 1 (1) | 7 (7)
Chills (General disorders) | 85 (97) | 90 (115)
Injection site erythema (General disorders) | 59 (82) | 57 (77)
Injection site pain (General disorders) | 204 (284) | 197 (272)
Injection site swelling (General disorders) | 38 (50) | 40 (55)
Pyrexia (General disorders) | 29 (34) | 40 (46)
Myalgia (Musculoskeletal and connective tissue disorders) | 153 (210) | 155 (214)
Headache (Nervous system disorders) | 119 (157) | 138 (182)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT05966090/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT05966090/SAP_001.pdf